CLINICAL TRIAL: NCT04613869
Title: Effects of Esketamine on Postoperative Pain, Anxiety and Depression in Patients Undergoing Tumor Surgery
Brief Title: The Effect of Esketamine on Patients Undergoing Tumor Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-818
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Tumor Surgery
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose esketamine group (Experimental): After the operation, 5 mg esketamine was injected intravenously for postoperative analgesia. PCIA formula: hydromorphone 6mg + esketamine 45mg + tropisetron 10mg into 0.9% sodium chloride injection 100ml, the first dose is 20ug/kg , Background dose 2ug/kg/h, single dose 4ug/kg/time
  Interventions: Drug: High-dose Esketamine hydrochloride+Hydromorphone
- Low-dose esketamine group (Experimental): After the operation, esketamine 2.5mg was injected intravenously for postoperative analgesia. PCIA formula: hydromorphone 6mg + esketamine 22.5mg + tropisetron 10mg into 0.9% sodium chloride injection 100ml, the first dose is 20ug/ kg, background dose 2ug/kg/h, single dose 4ug/kg/time
  Interventions: Drug: Low-dose Esketamine hydrochloride+Hydromorphone
- Control group (Placebo Comparator): PCIA formula: 6mg of hydromorphone + 10mg of tropisetron into 100ml of 0.9% sodium chloride injection, the first dose is 20ug/kg, the background dose is 2ug/kg/h, and the single dose is 4ug/kg/time.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: High-dose Esketamine hydrochloride+Hydromorphone — By adding different doses of esketamine to the postoperative analgesic pump, and the control group without adding this drug to observe the postoperative pain, anxiety and depression indicators of the surgical patients
  Arms: High-dose esketamine group
Drug: Low-dose Esketamine hydrochloride+Hydromorphone — By adding different doses of esketamine to the postoperative analgesic pump, and the control group without adding this drug to observe the postoperative pain, anxiety and depression indicators of the surgical patients
  Arms: Low-dose esketamine group
Drug: Hydromorphone — No esketamine added
  Arms: Control group

SUMMARY:
Although the acute and chronic postoperative pain of surgical patients has gradually been paid attention to, it has not yet been better resolved.and, the incidence of anxiety and depression in cancer patients is constantly increasing，The new analgesic anesthetic esketamine hydrochloride was launched in China last year，however, in the domestic and foreign literature, there are still few reports of esketamine hydrochloride in postoperative analgesia, and most of them are retrospective and small samples.This study aims to investigate whether esketamine has advantages over traditional opioids in terms of postoperative analgesia, anxiety and depression in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Patients undergoing elective tumor surgery
* Use intravenous analgesia pump (PCIA) after operation

Exclusion Criteria:

* Patients with severe infection or respiratory system diseases;
* Severe arrhythmia, unstable angina or myocardial infarction, heart failure;
* Patients with severe diseases of liver, kidney, endocrine or immune system; ·Patients with fever before operation;
* One month before operation Patients receiving chemotherapy, radiotherapy or immunotherapy;
* Drug or alcohol dependence;
* Mental illness, disturbance of consciousness and communication difficulties or inability to understand the questionnaire or refusal to complete;
* Long-term use of antidepressant and anxiety drugs;
* High intracranial pressure High intraocular pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate to severe pain | Within 72 hours after surgery
  Visual analog score is 4 points or more
Pain score | Within 72 hours after surgery
  Visual analog scale

SECONDARY OUTCOMES:
Adverse reactions | Within 72 hours after surgery
  Nausea, vomiting, lethargy, mental symptoms, etc.
Postoperative analgesia | Within 48 hours after surgery
  PCIA usage（ml）, PCIA compressions（frequency）, remedial analgesia measures（Name and dosage of intravenous analgesics）
Sedation | Within 48 hours after surgery
  Ramsay sedation score（The score is 1-6 points, the higher the score, the higher the degree of sedation, the ideal sedation score is 2 points）
Anxiety | Baseline (Before operation), 24 hours after operation, 72 hours after operation
  Hamilton Anxiety Scale（There are a total of 14 options. Each item is divided into 0-4 points according to the degree, and the score is 0-56 points. The total score is ≥29 points, which may be severe anxiety; ≥21 points, there must be obvious anxiety; ≥14 points, there must be Anxiety; more than 7 points, there may be anxiety; if less than 7, there are no anxiety symptoms.）
Depression | Baseline (Before operation), 24 hours after operation, 72 hours after operation
  Hamilton Depression Scale（There are a total of 17 options, and each item is divided into 0-4 points or 0-2 points according to the degree. The total score is less than 7 points: normal; the total score is 7~17 points: there may be depression; the total score is 17~24 points : There must be depression; total score> 24 points: severe depression）
Sleep condition | Within 72 hours after surgery
  Sleep quality（Self-assessment by the patient, the score is 1-5 points, the higher the score, the better the sleep）
Chronic pain | One month after surgery
  Chronic pain conversion rate（Follow-up one month after surgery, if there are still pain symptoms, it is chronic pain）

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Director — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No